CLINICAL TRIAL: NCT03109925
Title: Use of a Novel Radiopaque Embolic Agent in Prostatic Artery Embolisation for Symptomatic Benign Prostatic Enlargement
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHMRAD0042
Record Dates: First submitted 2017-03-13; First posted 2017-04-12 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: PAE; embolization; non-surgical; prostate artery embolization; radio-opaque embolic
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Single group of patients undergoing prostate artery embolization with a new embolic which is radio-opaque and can give a better idea of embolization distribution (DC Lumi Beads by BTG)
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radio-opaque embolic arm (Experimental): Patients will undergo intervention in the form of prostate artery embolization with the new radio-opaque embolic "Lumi-Bead" developed by BTG plc.
  Interventions: Device: DC Lumi Bead, BTG

INTERVENTIONS:
Device: DC Lumi Bead, BTG — Embolic agent which is radio-opaque

SUMMARY:
This is a study protocol for the use of a novel radiopaque embolic agent in the treatment of lower urinary tract Symptoms (LUTS) with prostatic artery embolisation (PAE). This study will allow us to evaluate the safety and efficacy of this embolic in PAE along with giving us a better understanding of embolic distribution.

DETAILED DESCRIPTION:
This is a study protocol for the use of a novel radiopaque embolic agent in the treatment of lower urinary tract Symptoms (LUTS) with prostatic artery embolisation (PAE). This study will allow us to evaluate the safety and efficacy of this embolic in PAE along with giving us a better understanding of embolic distribution. It would also give us answers to:

* How does embolic efficacy compare to current available embolic agents?
* Does enhancement on rotational CT correlate with embolic distribution?
* How does embolic distribution compare with tissue infarction?
* Does the density of embolic packing correlate with degree of infarction and volume loss?
* How predictable is superselective target embolisation?
* Does embolic distribution vary with anatomy and gland size?
* Does embolic distribution tally with glandular enhancement/ transitional zone vascularity?
* If visible, what is the effect and significance of non target embolisation? This is a cohort study aiming to recruit 22 patients to power a non-inferiority assessment comparing the novel embolic agent against current available embolics.

Data will be added to our on going local registry of patients who have undergone this procedure . This will provide information about how safe and effective it is for patients and how it compares to the other established embolic agents such as polyvinyl alcohol (PVA) and other spherical agents such as Embospheres and Embozenes.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-80 Moderate to severe lower urinary tract symptoms secondary to benign prostatic enlargement (BPE) IPSS>14, QOL≥4 Prostate volume ≥ 40 cc Maximum urinary flow rate < 12ml/s Medically refractory BPE > 6 months (or unable/ unwilling to tolerate medical treatment due to side effects)

Exclusion Criteria:

* Atherosclerosis of the prostatic arteries Surgical indications (Chronic retention, bladder diverticulae, urethral stenosis), detrusor instability, neurogenic bladder Malignancy (TRUS/ MRI/ Biopsy proven). PSA > 4 or high SWOP risk need prostate biopsy Urodynamics - non-obstructed eGFR ≤ 45ml min-1m-2

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2021-06-29 (Estimated); Study Completion 2021-06-29 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | 12 months
  Rate of adverse events compared with currently available other embolic agents

SECONDARY OUTCOMES:
Scale of symptomatic improvement | 12 months
  symptomatic improvement will be gauged used the internationally recognised IPSS questionnaire. Decrease in IPSS score in study participants will be compared against other embolic agents in the literature

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bryant, Principal Investigator — University of Hospital Southampton
Locations (1):
- Southampton General Hospital, University Hospital Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Currently there is no plan to make individual participant data available to other researchers.